CLINICAL TRIAL: NCT02783469
Title: Genetics of Diabetes Audit and Research in Tayside Scotland (DOLORisk Dundee)
Acronym: GoDARTS
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Collaborators: Wellcome Trust (Other); Diabetes UK (Other)
Responsible Party: Sponsor
Other Study IDs: 2003DM08
Record Dates: First submitted 2016-04-12; First posted 2016-05-26 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Neuropathic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for DNA/RNA Serum for biomarkers Urine for microalbumin, metabolites and proteins
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic neuropathic pain: Those with type 2 diabetes and painful neuropathy
  Interventions: Genetic: Identification of genetic causes of diabetic neuropathic pain
- Controls: Type 2 diabetics with non-painful neuropathy, or pain without neuropathy
  Interventions: Genetic: Identification of genetic causes of diabetic neuropathic pain

INTERVENTIONS:
Genetic: Identification of genetic causes of diabetic neuropathic pain

SUMMARY:
In 1997, the global prevalence of diabetes was estimated to be 125 million and this has risen to around 400 million in 2015. In addition diabetes has a number of complications including heart disease, blindness, kidney failure and amputation. This represents a significant burden on healthcare services. Type 2 diabetes (T2D) is caused by a combination of genetic and environmental factors. The aim of GoDARTS is to recruit participants with T2D to a registry to provide a platform with which to investigate the genetics of T2D, its complications and response to treatment. This study will investigate the genetic basis of diabetic neuropathic pain.

DETAILED DESCRIPTION:
GoDARTS is the genetics arm of the DARTS study, which was set up to identify all diabetes patients in the Tayside region. Its aim is to improve diabetes care over and above existing practices. Participants are invited to attend to provide blood samples for DNA/RNA analysis, provide baseline anthropometric, biochemical, blood pressure and heart rate measurements as well as completing a lifestyle questionnaire containing smoking, menopausal and physical activity items. Consent is also obtained to allow anonymous linkage to electronic medical records (EMR) through use of the Community Health Index (CHI) number, a unique patient identifier that is issued to everyone registered with a general practitioner in Scotland. GoDARTS is the first EMR linked cohort in the world and provides access to individual participant longitudinal data including biochemical, comorbidity and prescription records. These are live databases and are constantly being updated. This allows for the study of genetic factors influencing T2D, its comorbidities and response to therapy. Consent has also been obtained for re-contact by collaborators, allowing for further studies of related phenotypes to take place. One of these studies is DOLORisk Dundee which aims to identify genetic and environmental risk factors for neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation with GoDARTS
* Existing consent to be recontacted
* Identified as being currently alive
* Currently has a postal address
* age > 18 years
* Neuropathic

Exclusion Criteria:

* Unable to give consent
* No current postcode
* Identified as having died

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes patients and non-diabetic controls will be recruited from residents of the Tayside area of Scotland (n=411,749 according to SCI-Diabetes).
Sampling Method: Non-Probability Sample
Enrollment: 1915 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2009-05-31 (Actual); Study Completion 2009-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Palmer, PhD, Principal Investigator — University of Dundee
Locations (1):
- University of Dundee, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Morris AD, Boyle DI, MacAlpine R, Emslie-Smith A, Jung RT, Newton RW, MacDonald TM. The diabetes audit and research in Tayside Scotland (DARTS) study: electronic record linkage to create a diabetes register. DARTS/MEMO Collaboration. BMJ. 1997 Aug 30;315(7107):524-8. doi: 10.1136/bmj.315.7107.524. PMID 9329309
- [Result] Dujic T, Zhou K, Donnelly LA, Tavendale R, Palmer CN, Pearson ER. Association of Organic Cation Transporter 1 With Intolerance to Metformin in Type 2 Diabetes: A GoDARTS Study. Diabetes. 2015 May;64(5):1786-93. doi: 10.2337/db14-1388. Epub 2014 Dec 15. PMID 25510240
- [Result] Looker HC, Colombo M, Hess S, Brosnan MJ, Farran B, Dalton RN, Wong MC, Turner C, Palmer CN, Nogoceke E, Groop L, Salomaa V, Dunger DB, Agakov F, McKeigue PM, Colhoun HM; SUMMIT Investigators. Biomarkers of rapid chronic kidney disease progression in type 2 diabetes. Kidney Int. 2015 Oct;88(4):888-96. doi: 10.1038/ki.2015.199. Epub 2015 Jul 22. PMID 26200946
- [Result] Mahajan A, Sim X, Ng HJ, Manning A, Rivas MA, Highland HM, Locke AE, Grarup N, Im HK, Cingolani P, Flannick J, Fontanillas P, Fuchsberger C, Gaulton KJ, Teslovich TM, Rayner NW, Robertson NR, Beer NL, Rundle JK, Bork-Jensen J, Ladenvall C, Blancher C, Buck D, Buck G, Burtt NP, Gabriel S, Gjesing AP, Groves CJ, Hollensted M, Huyghe JR, Jackson AU, Jun G, Justesen JM, Mangino M, Murphy J, Neville M, Onofrio R, Small KS, Stringham HM, Syvanen AC, Trakalo J, Abecasis G, Bell GI, Blangero J, Cox NJ, Duggirala R, Hanis CL, Seielstad M, Wilson JG, Christensen C, Brandslund I, Rauramaa R, Surdulescu GL, Doney AS, Lannfelt L, Linneberg A, Isomaa B, Tuomi T, Jorgensen ME, Jorgensen T, Kuusisto J, Uusitupa M, Salomaa V, Spector TD, Morris AD, Palmer CN, Collins FS, Mohlke KL, Bergman RN, Ingelsson E, Lind L, Tuomilehto J, Hansen T, Watanabe RM, Prokopenko I, Dupuis J, Karpe F, Groop L, Laakso M, Pedersen O, Florez JC, Morris AP, Altshuler D, Meigs JB, Boehnke M, McCarthy MI, Lindgren CM, Gloyn AL; T2D-GENES consortium and GoT2D consortium. Identification and functional characterization of G6PC2 coding variants influencing glycemic traits define an effector transcript at the G6PC2-ABCB11 locus. PLoS Genet. 2015 Jan 27;11(1):e1004876. doi: 10.1371/journal.pgen.1004876. eCollection 2015 Jan. PMID 25625282
- [Result] Meng W, Deshmukh HA, Donnelly LA; Wellcome Trust Case Control Consortium 2 (WTCCC2); Surrogate markers for Micro- and Macro-vascular hard endpoints for Innovative diabetes Tools (SUMMIT) study group; Torrance N, Colhoun HM, Palmer CN, Smith BH. A Genome-wide Association Study Provides Evidence of Sex-specific Involvement of Chr1p35.1 (ZSCAN20-TLR12P) and Chr8p23.1 (HMGB1P46) With Diabetic Neuropathic Pain. EBioMedicine. 2015 Aug 4;2(10):1386-93. doi: 10.1016/j.ebiom.2015.08.001. eCollection 2015 Oct. PMID 26629533
- [Result] Meng W, Deshmukh HA, van Zuydam NR, Liu Y, Donnelly LA, Zhou K; Wellcome Trust Case Control Consortium 2 (WTCCC2); Surrogate Markers for Micro- and Macro-Vascular Hard Endpoints for Innovative Diabetes Tools (SUMMIT) Study Group; Morris AD, Colhoun HM, Palmer CN, Smith BH. A genome-wide association study suggests an association of Chr8p21.3 (GFRA2) with diabetic neuropathic pain. Eur J Pain. 2015 Mar;19(3):392-9. doi: 10.1002/ejp.560. PMID 24974787
- [Result] Mosley JD, Shaffer CM, Van Driest SL, Weeke PE, Wells QS, Karnes JH, Velez Edwards DR, Wei WQ, Teixeira PL, Bastarache L, Crawford DC, Li R, Manolio TA, Bottinger EP, McCarty CA, Linneman JG, Brilliant MH, Pacheco JA, Thompson W, Chisholm RL, Jarvik GP, Crosslin DR, Carrell DS, Baldwin E, Ralston J, Larson EB, Grafton J, Scrol A, Jouni H, Kullo IJ, Tromp G, Borthwick KM, Kuivaniemi H, Carey DJ, Ritchie MD, Bradford Y, Verma SS, Chute CG, Veluchamy A, Siddiqui MK, Palmer CN, Doney A, MahmoudPour SH, Maitland-van der Zee AH, Morris AD, Denny JC, Roden DM. A genome-wide association study identifies variants in KCNIP4 associated with ACE inhibitor-induced cough. Pharmacogenomics J. 2016 Jun;16(3):231-7. doi: 10.1038/tpj.2015.51. Epub 2015 Jul 14. PMID 26169577
- [Result] Postmus I, Trompet S, Deshmukh HA, Barnes MR, Li X, Warren HR, Chasman DI, Zhou K, Arsenault BJ, Donnelly LA, Wiggins KL, Avery CL, Griffin P, Feng Q, Taylor KD, Li G, Evans DS, Smith AV, de Keyser CE, Johnson AD, de Craen AJ, Stott DJ, Buckley BM, Ford I, Westendorp RG, Slagboom PE, Sattar N, Munroe PB, Sever P, Poulter N, Stanton A, Shields DC, O'Brien E, Shaw-Hawkins S, Chen YD, Nickerson DA, Smith JD, Dube MP, Boekholdt SM, Hovingh GK, Kastelein JJ, McKeigue PM, Betteridge J, Neil A, Durrington PN, Doney A, Carr F, Morris A, McCarthy MI, Groop L, Ahlqvist E; Welcome Trust Case Control Consortium; Bis JC, Rice K, Smith NL, Lumley T, Whitsel EA, Sturmer T, Boerwinkle E, Ngwa JS, O'Donnell CJ, Vasan RS, Wei WQ, Wilke RA, Liu CT, Sun F, Guo X, Heckbert SR, Post W, Sotoodehnia N, Arnold AM, Stafford JM, Ding J, Herrington DM, Kritchevsky SB, Eiriksdottir G, Launer LJ, Harris TB, Chu AY, Giulianini F, MacFadyen JG, Barratt BJ, Nyberg F, Stricker BH, Uitterlinden AG, Hofman A, Rivadeneira F, Emilsson V, Franco OH, Ridker PM, Gudnason V, Liu Y, Denny JC, Ballantyne CM, Rotter JI, Adrienne Cupples L, Psaty BM, Palmer CN, Tardif JC, Colhoun HM, Hitman G, Krauss RM, Wouter Jukema J, Caulfield MJ. Pharmacogenetic meta-analysis of genome-wide association studies of LDL cholesterol response to statins. Nat Commun. 2014 Oct 28;5:5068. doi: 10.1038/ncomms6068. PMID 25350695
- [Result] Zhou K, Donnelly L, Yang J, Li M, Deshmukh H, Van Zuydam N, Ahlqvist E; Wellcome Trust Case Control Consortium 2; Spencer CC, Groop L, Morris AD, Colhoun HM, Sham PC, McCarthy MI, Palmer CN, Pearson ER. Heritability of variation in glycaemic response to metformin: a genome-wide complex trait analysis. Lancet Diabetes Endocrinol. 2014 Jun;2(6):481-7. doi: 10.1016/S2213-8587(14)70050-6. Epub 2014 Mar 19. PMID 24731673
- [Result] Alkayyali S, Lajer M, Deshmukh H, Ahlqvist E, Colhoun H, Isomaa B, Rossing P, Groop L, Lyssenko V. Common variant in the HMGA2 gene increases susceptibility to nephropathy in patients with type 2 diabetes. Diabetologia. 2013 Feb;56(2):323-9. doi: 10.1007/s00125-012-2760-5. Epub 2012 Oct 31. PMID 23111731
- [Result] Deshmukh HA, Palmer CN, Morris AD, Colhoun HM. Investigation of known estimated glomerular filtration rate loci in patients with type 2 diabetes. Diabet Med. 2013 Oct;30(10):1230-5. doi: 10.1111/dme.12211. Epub 2013 May 14. PMID 23586973
- [Result] Donnelly LA, van Zuydam NR, Zhou K, Tavendale R, Carr F, Maitland-van der Zee AH, Leusink M, de Boer A, Doevendans PA, Asselbergs FW, Morris AD, Pearson ER, Klungel OH, Doney AS, Palmer CN. Robust association of the LPA locus with low-density lipoprotein cholesterol lowering response to statin treatment in a meta-analysis of 30 467 individuals from both randomized control trials and observational studies and association with coronary artery disease outcome during statin treatment. Pharmacogenet Genomics. 2013 Oct;23(10):518-25. doi: 10.1097/FPC.0b013e3283642fd6. PMID 23903772
- [Result] Liu Y, Wang M, Morris AD, Doney AS, Leese GP, Pearson ER, Palmer CN. Glycemic exposure and blood pressure influencing progression and remission of diabetic retinopathy: a longitudinal cohort study in GoDARTS. Diabetes Care. 2013 Dec;36(12):3979-84. doi: 10.2337/dc12-2392. Epub 2013 Oct 29. PMID 24170761
- [Result] Parry HM, Donnelly LA, Van Zuydam N, Doney AS, Elder DH, Morris AD, Struthers AD, Palmer CN, Lang CC; Wellcome Trust Case Control Consortium 2. Genetic variants predicting left ventricular hypertrophy in a diabetic population: a Go-DARTS study including meta-analysis. Cardiovasc Diabetol. 2013 Jul 23;12:109. doi: 10.1186/1475-2840-12-109. PMID 23879873
- [Result] Palmer CN, Maglio C, Pirazzi C, Burza MA, Adiels M, Burch L, Donnelly LA, Colhoun H, Doney AS, Dillon JF, Pearson ER, McCarthy M, Hattersley AT, Frayling T, Morris AD, Peltonen M, Svensson PA, Jacobson P, Boren J, Sjostrom L, Carlsson LM, Romeo S. Paradoxical lower serum triglyceride levels and higher type 2 diabetes mellitus susceptibility in obese individuals with the PNPLA3 148M variant. PLoS One. 2012;7(6):e39362. doi: 10.1371/journal.pone.0039362. Epub 2012 Jun 18. PMID 22724004
- [Result] Perry JR, Voight BF, Yengo L, Amin N, Dupuis J, Ganser M, Grallert H, Navarro P, Li M, Qi L, Steinthorsdottir V, Scott RA, Almgren P, Arking DE, Aulchenko Y, Balkau B, Benediktsson R, Bergman RN, Boerwinkle E, Bonnycastle L, Burtt NP, Campbell H, Charpentier G, Collins FS, Gieger C, Green T, Hadjadj S, Hattersley AT, Herder C, Hofman A, Johnson AD, Kottgen A, Kraft P, Labrune Y, Langenberg C, Manning AK, Mohlke KL, Morris AP, Oostra B, Pankow J, Petersen AK, Pramstaller PP, Prokopenko I, Rathmann W, Rayner W, Roden M, Rudan I, Rybin D, Scott LJ, Sigurdsson G, Sladek R, Thorleifsson G, Thorsteinsdottir U, Tuomilehto J, Uitterlinden AG, Vivequin S, Weedon MN, Wright AF; MAGIC; DIAGRAM Consortium; GIANT Consortium; Hu FB, Illig T, Kao L, Meigs JB, Wilson JF, Stefansson K, van Duijn C, Altschuler D, Morris AD, Boehnke M, McCarthy MI, Froguel P, Palmer CN, Wareham NJ, Groop L, Frayling TM, Cauchi S. Stratifying type 2 diabetes cases by BMI identifies genetic risk variants in LAMA1 and enrichment for risk variants in lean compared to obese cases. PLoS Genet. 2012 May;8(5):e1002741. doi: 10.1371/journal.pgen.1002741. Epub 2012 May 31. PMID 22693455
- [Result] Warren LL, Li L, Nelson MR, Ehm MG, Shen J, Fraser DJ, Aponte JL, Nangle KL, Slater AJ, Woollard PM, Hall MD, Topp SD, Yuan X, Cardon LR, Chissoe SL, Mooser V, Morris AD, Palmer CN, Perry JR, Frayling TM, Whittaker JC, Waterworth DM. Deep resequencing unveils genetic architecture of ADIPOQ and identifies a novel low-frequency variant strongly associated with adiponectin variation. Diabetes. 2012 May;61(5):1297-301. doi: 10.2337/db11-0985. Epub 2012 Mar 8. PMID 22403302
- [Result] Donnelly LA, Doney AS, Tavendale R, Lang CC, Pearson ER, Colhoun HM, McCarthy MI, Hattersley AT, Morris AD, Palmer CN. Common nonsynonymous substitutions in SLCO1B1 predispose to statin intolerance in routinely treated individuals with type 2 diabetes: a go-DARTS study. Clin Pharmacol Ther. 2011 Feb;89(2):210-6. doi: 10.1038/clpt.2010.255. Epub 2010 Dec 22. PMID 21178985
- [Result] GoDARTS and UKPDS Diabetes Pharmacogenetics Study Group; Wellcome Trust Case Control Consortium 2; Zhou K, Bellenguez C, Spencer CC, Bennett AJ, Coleman RL, Tavendale R, Hawley SA, Donnelly LA, Schofield C, Groves CJ, Burch L, Carr F, Strange A, Freeman C, Blackwell JM, Bramon E, Brown MA, Casas JP, Corvin A, Craddock N, Deloukas P, Dronov S, Duncanson A, Edkins S, Gray E, Hunt S, Jankowski J, Langford C, Markus HS, Mathew CG, Plomin R, Rautanen A, Sawcer SJ, Samani NJ, Trembath R, Viswanathan AC, Wood NW; MAGIC investigators; Harries LW, Hattersley AT, Doney AS, Colhoun H, Morris AD, Sutherland C, Hardie DG, Peltonen L, McCarthy MI, Holman RR, Palmer CN, Donnelly P, Pearson ER. Common variants near ATM are associated with glycemic response to metformin in type 2 diabetes. Nat Genet. 2011 Feb;43(2):117-20. doi: 10.1038/ng.735. Epub 2010 Dec 26. PMID 21186350
- [Result] Grant RW, Wexler DJ. Loss-of-function CYP2C9 variants: finding the correct clinical role for Type 2 diabetes pharmacogenetic testing. Expert Rev Cardiovasc Ther. 2010 Mar;8(3):339-43. doi: 10.1586/erc.10.5. PMID 20222813
- [Result] Palmer CN, Kimber CH, Doney AS, Proia AS, Morris AD, Gaetani E, Quarta M, Smith RC, Pola R. Combined effect of inflammatory gene polymorphisms and the risk of ischemic stroke in a prospective cohort of subjects with type 2 diabetes: a Go-DARTS study. Diabetes. 2010 Nov;59(11):2945-8. doi: 10.2337/db09-1690. Epub 2010 Jul 9. PMID 20622166
- [Result] Zhou K, Donnelly L, Burch L, Tavendale R, Doney AS, Leese G, Hattersley AT, McCarthy MI, Morris AD, Lang CC, Palmer CN, Pearson ER. Loss-of-function CYP2C9 variants improve therapeutic response to sulfonylureas in type 2 diabetes: a Go-DARTS study. Clin Pharmacol Ther. 2010 Jan;87(1):52-6. doi: 10.1038/clpt.2009.176. Epub 2009 Sep 30. PMID 19794412
- [Result] Doney AS, Leese GP, Olson J, Morris AD, Palmer CN. The Y402H variant of complement factor H is associated with age-related macular degeneration but not with diabetic retinal disease in the Go-DARTS study. Diabet Med. 2009 May;26(5):460-5. doi: 10.1111/j.1464-5491.2009.02719.x. PMID 19646183
- [Result] Doney AS, Dannfald J, Kimber CH, Donnelly LA, Pearson E, Morris AD, Palmer CN. The FTO gene is associated with an atherogenic lipid profile and myocardial infarction in patients with type 2 diabetes: a Genetics of Diabetes Audit and Research Study in Tayside Scotland (Go-DARTS) study. Circ Cardiovasc Genet. 2009 Jun;2(3):255-9. doi: 10.1161/CIRCGENETICS.108.822320. Epub 2009 Mar 30. PMID 20031593
- [Result] Zhou K, Donnelly LA, Kimber CH, Donnan PT, Doney AS, Leese G, Hattersley AT, McCarthy MI, Morris AD, Palmer CN, Pearson ER. Reduced-function SLC22A1 polymorphisms encoding organic cation transporter 1 and glycemic response to metformin: a GoDARTS study. Diabetes. 2009 Jun;58(6):1434-9. doi: 10.2337/db08-0896. Epub 2009 Mar 31. PMID 19336679
- [Result] Donnelly LA, Doney AS, Dannfald J, Whitley AL, Lang CC, Morris AD, Donnan PT, Palmer CN. A paucimorphic variant in the HMG-CoA reductase gene is associated with lipid-lowering response to statin treatment in diabetes: a GoDARTS study. Pharmacogenet Genomics. 2008 Dec;18(12):1021-6. doi: 10.1097/FPC.0b013e3283106071. PMID 18815589
- [Result] Donnelly LA, Palmer CN, Whitley AL, Lang CC, Doney AS, Morris AD, Donnan PT. Apolipoprotein E genotypes are associated with lipid-lowering responses to statin treatment in diabetes: a Go-DARTS study. Pharmacogenet Genomics. 2008 Apr;18(4):279-87. doi: 10.1097/FPC.0b013e3282f60aad. PMID 18334912
- [Result] Vitart V, Rudan I, Hayward C, Gray NK, Floyd J, Palmer CN, Knott SA, Kolcic I, Polasek O, Graessler J, Wilson JF, Marinaki A, Riches PL, Shu X, Janicijevic B, Smolej-Narancic N, Gorgoni B, Morgan J, Campbell S, Biloglav Z, Barac-Lauc L, Pericic M, Klaric IM, Zgaga L, Skaric-Juric T, Wild SH, Richardson WA, Hohenstein P, Kimber CH, Tenesa A, Donnelly LA, Fairbanks LD, Aringer M, McKeigue PM, Ralston SH, Morris AD, Rudan P, Hastie ND, Campbell H, Wright AF. SLC2A9 is a newly identified urate transporter influencing serum urate concentration, urate excretion and gout. Nat Genet. 2008 Apr;40(4):437-42. doi: 10.1038/ng.106. Epub 2008 Mar 9. PMID 18327257
- [Result] Gudmundsson J, Sulem P, Steinthorsdottir V, Bergthorsson JT, Thorleifsson G, Manolescu A, Rafnar T, Gudbjartsson D, Agnarsson BA, Baker A, Sigurdsson A, Benediktsdottir KR, Jakobsdottir M, Blondal T, Stacey SN, Helgason A, Gunnarsdottir S, Olafsdottir A, Kristinsson KT, Birgisdottir B, Ghosh S, Thorlacius S, Magnusdottir D, Stefansdottir G, Kristjansson K, Bagger Y, Wilensky RL, Reilly MP, Morris AD, Kimber CH, Adeyemo A, Chen Y, Zhou J, So WY, Tong PC, Ng MC, Hansen T, Andersen G, Borch-Johnsen K, Jorgensen T, Tres A, Fuertes F, Ruiz-Echarri M, Asin L, Saez B, van Boven E, Klaver S, Swinkels DW, Aben KK, Graif T, Cashy J, Suarez BK, van Vierssen Trip O, Frigge ML, Ober C, Hofker MH, Wijmenga C, Christiansen C, Rader DJ, Palmer CN, Rotimi C, Chan JC, Pedersen O, Sigurdsson G, Benediktsson R, Jonsson E, Einarsson GV, Mayordomo JI, Catalona WJ, Kiemeney LA, Barkardottir RB, Gulcher JR, Thorsteinsdottir U, Kong A, Stefansson K. Two variants on chromosome 17 confer prostate cancer risk, and the one in TCF2 protects against type 2 diabetes. Nat Genet. 2007 Aug;39(8):977-83. doi: 10.1038/ng2062. Epub 2007 Jul 1. PMID 17603485
- [Result] Kimber CH, Doney AS, Pearson ER, McCarthy MI, Hattersley AT, Leese GP, Morris AD, Palmer CN. TCF7L2 in the Go-DARTS study: evidence for a gene dose effect on both diabetes susceptibility and control of glucose levels. Diabetologia. 2007 Jun;50(6):1186-91. doi: 10.1007/s00125-007-0661-9. Epub 2007 Apr 11. PMID 17429603
- [Result] Pearson ER, Donnelly LA, Kimber C, Whitley A, Doney AS, McCarthy MI, Hattersley AT, Morris AD, Palmer CN. Variation in TCF7L2 influences therapeutic response to sulfonylureas: a GoDARTs study. Diabetes. 2007 Aug;56(8):2178-82. doi: 10.2337/db07-0440. Epub 2007 May 22. PMID 17519421
- [Result] Sandhu MS, Weedon MN, Fawcett KA, Wasson J, Debenham SL, Daly A, Lango H, Frayling TM, Neumann RJ, Sherva R, Blech I, Pharoah PD, Palmer CN, Kimber C, Tavendale R, Morris AD, McCarthy MI, Walker M, Hitman G, Glaser B, Permutt MA, Hattersley AT, Wareham NJ, Barroso I. Common variants in WFS1 confer risk of type 2 diabetes. Nat Genet. 2007 Aug;39(8):951-3. doi: 10.1038/ng2067. Epub 2007 Jul 1. PMID 17603484
- [Result] Doney AS, Fischer B, Lee SP, Morris AD, Leese G, Palmer CN. Association of common variation in the PPARA gene with incident myocardial infarction in individuals with type 2 diabetes: a Go-DARTS study. Nucl Recept. 2005 Nov 25;3:4. doi: 10.1186/1478-1336-3-4. PMID 16309557
- [Result] Doney AS, Lee S, Leese GP, Morris AD, Palmer CN. Increased cardiovascular morbidity and mortality in type 2 diabetes is associated with the glutathione S transferase theta-null genotype: a Go-DARTS study. Circulation. 2005 Jun 7;111(22):2927-34. doi: 10.1161/CIRCULATIONAHA.104.509224. Epub 2005 May 31. PMID 15927971
- [Result] Doney AS, Fischer B, Leese G, Morris AD, Palmer CN. Cardiovascular risk in type 2 diabetes is associated with variation at the PPARG locus: a Go-DARTS study. Arterioscler Thromb Vasc Biol. 2004 Dec;24(12):2403-7. doi: 10.1161/01.ATV.0000147897.57527.e4. Epub 2004 Oct 14. PMID 15486307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At baseline recruitment, participants of GoDARTS who had provided consent to be contacted about related studies, were sent and invited to complete and return a DOLORisk Dundee questionnaire on neuropathic pain and pain-related traits, between December 2016. Approximately 18 months later, participants of the baseline survey who provided further consent to be recontacted, were sent a similar follow-up questionnaire.
Groups:
- GoDARTS: Participants of the baseline DOLORisk Dundee survey
Period: Overall Study
Arm/Group | GoDARTS
Started | 1915
Completed | 1915
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who returned a completed DOLORisk Dundee questionnaire during the baseline survey
Groups:
- GoDARTS: Participants of the DOLORisk Dundee baseline survey
Arm/Group | GoDARTS
Number analyzed (Participants) | 1915
Age, Categorical [Count of Participants; unit: Participants] — Population: Age data is missing for 3 participants
  Participants
    number analyzed (Participants) | 1912
    <=18 years | 0
    Between 18 and 65 years | 491
    >=65 years | 1421
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Age data is missing for 3 participants
  years
    number analyzed (Participants) | 1912
    (all) | 71 [64 to 77]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data is missing for 3 participants
  Participants
    number analyzed (Participants) | 1912
    Female | 754
    Male | 1158
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1904
  More than one race | 0
  Unknown or Not Reported | 11
Douleur Neuropathique en Quatre Questions (DN4) [Count of Participants; unit: Participants] — The self-report version of the Douleur Neuropathique en Quatre Questions (DN4) is a validated screening tool for neuropathic pain (suitable for use in online and postal surveys). It consists of seven questions relating to the quality and sensation of pain experienced by the participant (burning, painful cold, electric shocks, tingling, pins and needles, numbness, and itching). Each question has a yes/no response with each 'yes' response scoring 1 and 'no' scoring 0. Scores of ≥3/7 suggest pain of neuropathic characteristics. Population: Only people who reported current pain or currently taking pain medication were asked to complete the DN4 (n=1276). Participants are only included in the DN4 count if all items in the DN4 are non-missing (n=875).
  Participants
    number analyzed (Participants) | 875
    DN4 ≥ 3 | 348
    DN4 < 3 | 527
Pain Duration [Count of Participants; unit: Participants] — Population: Only participants who reported current pain or currently taking pain medication were asked to complete the pain duration question (n=1276). Pain duration is missing for 38 of these participants (n=1238).
  Participants
    number analyzed (Participants) | 1238
    Duration ≥ 3 months | 1144
    Duration < 3 months | 94

OUTCOME MEASURES:

1. Primary Outcome: Neuropathic Pain
Description: Neuropathic pain will be identified according to the validated Douleur Neuropathique en Quatre Questions (DN4) questionnaire (English language)
Time Frame: April 2016 - December 2016
Population: Chronic neuropathic pain = DN4 ≥ 3 & pain duration ≥ 3 months Chronic nociceptive pain = DN4 < 3 & pain duration ≥ 3 months No pain = no current pain or currently taking pain medication
  Note: Participants were included in the chronic neuropathic pain group if they satisfied the above criteria, regardless of the number of missing DN4 items, and excluded from the chronic nociceptive pain group if the number of missing DN4 items plus the their DN4 score totalled 3 or more.
Measure: Count of Participants; unit: Participants
Arm/Group | GoDARTS
Number analyzed (Participants) | 1503
Participants
  Chronic Neuropathic Pain | 482
  Chronic Nociceptive Pain | 461
  No Pain | 560

ADVERSE EVENTS:
Arm/Group | GoDARTS
Serious Adverse Events (participants affected / at risk) | 0/1915
Other Adverse Events (participants affected / at risk) | 0/1915

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes